CLINICAL TRIAL: NCT01462448
Title: Study to Identify the Genetic Variations Associated With Phantom Limb Pain
Status: Completed | Type: Observational
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 20429; HU0001-11-1-0005 (Other Grant/Funding Number: Uniformed Services University of Health Sciences (USUHS))
Record Dates: First submitted 2011-10-24; First posted 2011-10-31 (Estimated); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Phantom Limb
Keywords: Phantom Limb; Genetic Variation; DNA Sequence Analysis; Amputation, Traumatic; Single Nucleotide Polymorphism; Visual Analog Pain Scale; Brain-Derived Neurotrophic Factor; Inflammatory Antibody; Peripheral Nerve Damage
MeSH Terms: conditions — Phantom Limb; Amputation, Traumatic; Neuritis | interventions — Blood Specimen Collection; Phlebotomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Phantom Limb Pain: Subjects will have lower or upper extremity amputation(s) that have resulted in the presence of phantom limb pain.
  Interventions: Procedure: Blood Draw
- No Phantom Limb Pain: Subjects in the group will have a lower or upper extremity amputation(s) without the presence of phantom limb sensation.
  Interventions: Procedure: Blood Draw

INTERVENTIONS:
Procedure: Blood Draw — Single blood draw of 30 ml
  Other Names: Venipuncture

SUMMARY:
The purpose of this study is to determine if there is a genetic component to phantom limb pain. DNA will be analyzed for single nucleotide polymorphisms (SNPs) between the control and phantom limb pain group. Total RNA will also be isolated and profiled to asses the degree to which our gene(s) of interest are expressed in the presence or absence of phantom limb pain. Some proteins, such as inflammatory antibodies or the neurotrophin brain-derived neurotrophic factor (BDNF), will also be assessed for their association(s) with phantom limb pain.

DETAILED DESCRIPTION:
Most patients (90-95%)with major limb amputations experience a phantom limb--the vivid impression that the limb is still present. In many cases, the sensation is painful for reasons that are currently not well understood. A small subset of amputees (<10%) never experience phantom limb pain (PLP), the painful sensation felt in the amputated limb. This difference suggests that there may be a genetic component that precludes some patients from ever experiencing PLP. Understanding the genetic components of PLP may help in predicting which patients will experience PLP and which amputees will respond to the various treatment options available.

In order to understand the genetic aspects and ultimately develop more effective treatment options in the future, patients with and without PLP will be asked to give 30 mls of blood after overnight fasting. These blood samples will be de-identified and sent to the National Institutes of Health (NIH) in Bethesda, Maryland, where all of the genetic analyses will take place.

ELIGIBILITY:
Chronic PLP Group:

* At least 18 years of age.
* Written informed consent and written authorization for use or release of health and research study information
* Single or multiple upper and/or lower limb amputation
* At least three months post-amputation
* Ability to follow study instructions and likely to complete required visit(s)
* Experienced PLP for at least one month and at least 3 times per week
* Phantom limb pain differentiated from residual limb pain by physical exam.
* Subjects taking blood thinners or other medications that do not increase risk during a blood draw.

Non-Chronic PLP Group:

* At least 18 years of age.
* Written informed consent and written authorization for use or release of health and research study information
* Single or multiple upper and/or lower limb(s) amputation
* At least three months post-amputation
* Ability to follow study instructions and likely to complete required visit(s)
* Experienced PLP less than 10 times total and/or for less than two weeks
* Subjects taking blood thinners or other medications that do not increase risk during a blood draw.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects to be recruited at WRNMMC will be military health care beneficiaries age 18 and older who have sustained one or more amputations.
Sampling Method: Non-Probability Sample
Enrollment: 726 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2023-08-06 (Actual)

PRIMARY OUTCOMES:
Identification of Unique Single Nucleotides Polymorphisms (SNPs) associated with Phantom Limb Pain (PLP) | 5 years
  The primary outcome measure for this study is the identification of unique SNPs that may correlate with PLP. Patients will undergo a one-time blood draw and fill out a survey characterizing their phantom limb pain. The PLP characteristics along with DNA analysis using Affymetrix SNP chip technology will be used to match genotype with phenotype.

SECONDARY OUTCOMES:
Correlation between Phantom Limb Pain (PLP) and Blood Levels of Antibodies Associated with Peripheral Nerve Damage | 5 years
  The underlying hypothesis of the secondary outcome measure is that damage to peripheral nerves provokes a humoral immune response to neuronal and glial proteins that can be detected by measuring specific antibodies in blood. The data obtained will lead to a more complete understanding of pathogenic mechanisms in PLP and potential biomarkers for sub-classification, prognosis, and intervention.
Correlation between Phantom Limb Pain (PLP) and Serum Levels of Brain-derived Neurotrophic Factor (BDNF) | 5 years
  BDNF has been implicated in pain nociception and is therefore pertinent to our study of phantom limb pain. After peripheral nerve injury, BDNF expression is dramatically increased in pain receptors of the brainstem.
Correlation between Phantom Limb Pain (PLP) and Unique Transcribed RNA | 5 years
  Many underlying causes for neuropathic pain involve changes in messenger ribonucleic acid (mRNA) levels because of altered gene expression or transcript stability. The study will isolate total RNA from blood and measure the relative amounts of transcribed RNA under the condition of phantom limb pain or no phantom limb pain.

CONTACTS AND LOCATIONS:
Overall Officials: Paul F. Pasquina, MD, MC, Principal Investigator — Walter Reed National Military Medical Center (WRNMMC)
Locations (1):
- Walter Reed National Military Medical Center (WRNMMC), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montoya P, Larbig W, Grulke N, Flor H, Taub E, Birbaumer N. The relationship of phantom limb pain to other phantom limb phenomena in upper extremity amputees. Pain. 1997 Aug;72(1-2):87-93. doi: 10.1016/s0304-3959(97)00004-3. PMID 9272791
- [Background] Kooijman CM, Dijkstra PU, Geertzen JHB, Elzinga A, van der Schans CP. Phantom pain and phantom sensations in upper limb amputees: an epidemiological study. Pain. 2000 Jul;87(1):33-41. doi: 10.1016/S0304-3959(00)00264-5. PMID 10863043
- [Background] Ramachandran VS, Hirstein W. The perception of phantom limbs. The D. O. Hebb lecture. Brain. 1998 Sep;121 ( Pt 9):1603-30. doi: 10.1093/brain/121.9.1603. PMID 9762952
- [Background] Sherman RA, Sherman CJ, Parker L. Chronic phantom and stump pain among American veterans: results of a survey. Pain. 1984 Jan;18(1):83-95. doi: 10.1016/0304-3959(84)90128-3. PMID 6709380
- [Background] Katz J, Melzack R. Pain 'memories' in phantom limbs: review and clinical observations. Pain. 1990 Dec;43(3):319-336. doi: 10.1016/0304-3959(90)90029-D. PMID 2293143
- [Background] Jensen TS, Krebs B, Nielsen J, Rasmussen P. Phantom limb, phantom pain and stump pain in amputees during the first 6 months following limb amputation. Pain. 1983 Nov;17(3):243-256. doi: 10.1016/0304-3959(83)90097-0. PMID 6657285